CLINICAL TRIAL: NCT06343285
Title: Upper Limb Tremor Reduction in Essential Tremor Patients
Acronym: ULTRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Encora, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20231215
Record Dates: First submitted 2024-01-26; First posted 2024-04-02 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Intervention Model Description: Three different arms in a randomized order
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization schedule maintained by non-Clinical personnel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Arm 1 (Sham Comparator): Inactive stimulation - device is powered on, but motors are inactive and amplitude is set to 0%
  Interventions: Device: Encora Therapeutics Tremor Reduction Device
- Arm 2 (Active Comparator): Treatment with the wearable device set to a specific dermatome, duty cycle and amplitude
  Interventions: Device: Encora Therapeutics Tremor Reduction Device
- Arm 3 (Active Comparator): treatment with the wearable device set to frequency-match the subject's tremor, duty cycle of and amplitude are set
  Interventions: Device: Encora Therapeutics Tremor Reduction Device

INTERVENTIONS:
Device: Encora Therapeutics Tremor Reduction Device — The proposed therapeutic device uses vibration motors positioned around the wrist that provide on-demand-therapy to suppress resting, postural, or action tremors of the hand.

SUMMARY:
This study is designed to demonstrate the safety, tolerability, and efficacy of the Encora Therapeutics Tremor Mitigation Device in subjects with upper limb tremor caused by Essential Tremor.

DETAILED DESCRIPTION:
A prospective, randomized, blinded clinical trial. Subjects meeting all inclusion criteria will have five days of treatment with each of the three arms, received in a randomized order. Subjects will complete two rounds of assessments each day.

Arm 1: Inactive stim Arm 2: Stim therapy utilizing a specific dermatome Arm 3: Stim therapy utilizing a tailored frequency

ELIGIBILITY:
Inclusion/Exclusion:

Inclusion Criteria:

1. Between the ages of 22 and 80 years of age
2. A diagnosis of essential tremor (definite or probable based on TRIG criteria)
3. At least one hand exhibiting tremor > 2 as assessed by the Essential Tremor Rating
4. Assessment Scale (TETRAS) finger to nose task, duck wing task, OR Archimedes Spiral completed during the Screening visit
5. Stable tremor medications for at least 30 days prior to enrollment and the ability to maintain stable medications through the duration of the study

Randomization Inclusion Criteria

1. During the Baseline evaluation period, a median tremor score of > 2 on at least one hand as assessed by the TETRAS finger to nose task, the duck wing task, OR the Archimedes Spiral AND
2. During the Baseline evaluation period, a median score of > 3 on any one of the subject-assessed items of the Bain & Findley Activities of Daily Living Scale (BF-ADL)

Exclusion Criteria:

1. Previous surgical interventions for tremor reduction on the upper limb being used for inclusion in this study (eg, thalamotomy procedure, including Stereotactic Thalamotomy, Gamma Knife Radiosurgical Thalamotomy, or focused ultrasound)
2. Use of botulinum toxin for treatment to hand tremor within six months of enrollment
3. Suspected or diagnosed epilepsy or other seizure disorder
4. Other possible causes of tremor, including Parkinson's disease, drug-induced tremor, or dystonia
5. Pregnant
6. Swollen, infected, inflamed areas, or skin eruptions, open wounds, or cancerous lesions of skin at stimulation site
7. Numbness, tingling or pain affecting the tested upper extremity (eg, suspected or confirmed peripheral neuropathy, carpal tunnel syndrome)
8. Known allergy to silicone
9. Subjects are unable or unwilling to comply with the protocol requirements
10. Subject is part of a vulnerable population who is unable to give Informed Consent for reasons of incapacity, dementia, immaturity, adverse personal circumstances or lack of autonomy. This may include individuals with mental disability, persons in nursing homes, children, impoverished persons, persons in emergency situations, homeless persons, nomads, refugees, and those incapable of giving informed consent.
11. Vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces, and persons kept in detention.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Tolerability (Rate of Subject-Assessed Comfort with Stimulation) | At the end of the 5-day treatment period in all randomization arms
  The rate of subject-assessed comfort with stimulation, on a Subject Stimulation Tolerance Questionnaire as measured by % of patient who tolerated the treatment either none of the time, some of the time or all of the time.
Safety (Rate of Adverse Events) | At the end of the 5-day treatment period in all randomization arms
  The rate of occurrence of adverse events (AEs) as both total numbers of AEs experienced throughout the study and percentage of subjects who experienced an AE.

SECONDARY OUTCOMES:
Bain & Findley Activity of Daily Living (BF-ADL) #2 | At the end of the 5-day treatment period in all randomization arms
  Use a spoon to drink soup: assess ability to perform task, score ranges from 1 (without difficulty) to 4 (cannot do by yourself).
BF-ADL #4 | At the end of the 5-day treatment period in all randomization arms
  Pour milk from a carton: assess ability to perform task, score ranges from 1 (without difficulty) to 4 (cannot do by yourself).
BF-ADL #17 | At the end of the 5-day treatment period in all randomization arms
  Dial a telephone: assess ability to perform task, score ranges from 1 (without difficulty) to 4 (cannot do by yourself).
BF-ADL #21 | At the end of the 5-day treatment period in all randomization arms
  Insert an electric plug into a socket: assess ability to perform task, score ranges from 1 (without difficulty) to 4 (cannot do by yourself).
Patient Global Impression of Change (PGI-C) | At the end of the 5-day treatment period in all randomization arms
  Measures change in condition as compared to baseline, score ranges from 1 = Very much improved to 7 = Very much worse.
Clinician Global Impression of Change (CGI-C) | At the end of the 5-day treatment period in all randomization arms
  Measures change in condition as compared to baseline, score ranges from 1 = Very much improved to 7 = Very much worse.
Tremor power as measured by gyroscope | At the end of the 5-day treatment period in all randomization arms
  Objective, sensor-based metric for tremor measurement.

OTHER OUTCOMES:
The Essential Tremor Rating Scale (TETRAS) #2.4 | At the end of the 5-day treatment period in all randomization arms
  The performance section of TETRAS has 9 items rated 0-4 and a maximum total score of 64. Item 4 is comprised of 3 tasks (Extended Arm, Duck Wing, Finger-to-Nose) related to upper limb tremor, with a score ranging from 0-12.
TETRAS #2.6 | At the end of the 5-day treatment period in all randomization arms
  The performance section of TETRAS has 9 items rated 0-4 and a maximum total score of 64. Item 6 is the Archimedes Spiral task, with a score ranging from 0-4.
TETRAS #2.8 | At the end of the 5-day treatment period in all randomization arms
  The performance section of TETRAS has 9 items rated 0-4 and a maximum total score of 64. Item 6 is the Dot Approximation task, with a score ranging from 0-4.
Patient Global Impression of Severity (PGI-S) | At the end of the 5-day treatment period in all randomization arms
  Rating of condition severity in the past week, with score ranges from 1 = Minimal to 5 = Very Severe.
Clinician Global Impression of Severity (CGI-S) | At the end of the 5-day treatment period in all randomization arms
  Rating of condition severity in the past week, with score ranges from 1 = Minimal to 5 = Very Severe.
Tremor power as measured by accelerometer | At the end of the 5-day treatment period in all randomization arms
  Objective, sensor-based metric for tremor measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Kristi Winterfeldt, MSHS, Principal Investigator — Encora Therapeutics
Locations (1):
- Encora Therapeutics, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No